CLINICAL TRIAL: NCT00493064
Title: Niacin (as a Vasodilator), and a Topical Steroid (for Macular Edema), Non-Ischemic CRVO,HRVO,BRVO
Brief Title: To Study the Effectiveness and Safety of Niacin and a Topical Steroid Eye Drop to Treat Retinal Vein Occlusions
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-21
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Niacin; prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective active treatment (Experimental): Niacin 500mg TID PO for treatment of retinal vein occlusions.
  Interventions: Drug: Nicotinic acid; Drug: Prednisolone acetate

INTERVENTIONS:
Drug: Nicotinic acid — topical eye drops
  Other Names: Niacin
Drug: Prednisolone acetate — topical eye drops

SUMMARY:
The purpose of this study is to determine whether Niacin, a B vitamin, may act as a vasodilator to encourage earlier formation of collateral blood vessels that may serve to bypass the obstructed vein in the eye. The topical steroid eye drops are aimed at reducing swelling in the retina, until the collateral vessels have a chance to develop.

DETAILED DESCRIPTION:
The aim of this study is to develop a less risky, yet effective and more sustainable treatment for retinal vein occlusions than the current commonly used approach of repeated intravitreal triamcinolone acetonide (Kenalog) injections. The types of retinal vein occlusion that are being studied include central (CRVO), hemi-retinal (HRVO), and branch (BRVO) retinal vein occlusion. Niacin, (Nicotinic Acid, not Nicotinamide)a B-vitamin, has lipid lowering and vasodilating properties. The combination of Niacin and Prednisolone Acetate steroid eye drops as a non-invasive treatment approach was developed by the Principal Investigator. The Niacin dilates the retinal vessels, hopefully encouraging earlier collateral vessel formation aimed at bypassing the venous obstruction, thus restoring venous outflow. The Prednisolone Acetate steroid eye drops are aimed at reducing vascular leakage and therefore the macular edema in the eye while the Niacin is taking effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand the study procedures, agree to participate, and give written consent.
* Patient must have central retinal vein occlusion, hemi-retinal vein occlusion or branch retinal vein occlusion.
* Patients must be able to follow the study medication regimen.
* Patients must agree to return for the once monthly eye exams.
* Patients must agree to have liver function tests performed on a regular basis.
* Patients must agree to have regular appointments with their Internist on an established basis.

Exclusion Criteria:

* Patients with active Gout, or high levels of Uric
* Patients may not be pregnant or lactating.
* The Principal Investigator reserves the right to exclude any patient who he feels will not make a good candidate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gaynon, MD, Principal Investigator — Palo Alto Medical Foundation
Locations (1):
- Palo Alto Medical Foundation Department of Ophthalmology, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Active Treatment
Started | 63
Completed | 52
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Prospective Active Treatment
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With An Improvement in Vision, as Measured by an Increase of 15 Letters on the Early Treatment Diabetic Retinopathy Study (EDTRS) Vision Chart.
Description: improvement with combination of niacin and topical prednisolone acetate
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Active Treatment
Number analyzed (Participants) | 63
Participants | 63

2. Secondary Outcome: A Decrease in the Thickness of the Retina
Description: data not available
Time Frame: one year
Population: Although data for this outcome measure was collected, however, data are not available. The PI is retired and no longer works in the organization. Sincere efforts were made to obtain the data, however, no data are available for this outcome.
Arm/Group | Prospective Active Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No information regarding the Adverse Events is available. The PI is retired and no longer works for the organization. Sincere efforts were made to obtain the data, however, no Adverse Events data are available.
Arm/Group | Prospective Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No